CLINICAL TRIAL: NCT03689764
Title: Effects of Interactive Video Game-based Exercise on Balance of Persons With Parkinson's Disease
Brief Title: Video Game-based Exercise for Persons With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Lai chien hung, Professor, Taipei Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 201311032
Record Dates: First submitted 2018-09-24; First posted 2018-09-28 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A underwent interactive video game-based exercise for the initial 6 weeks, with no treatment in the subsequent 6 weeks. The exercise program consisted of 30-minute sessions 3 times per week for 6 weeks. Outcomes were measured at weeks 0, 6, and 12.
  Interventions: Other: interactive video game-based exercise; Other: no intervention
- Group B (Experimental): Group B had no intervention in the first 6 weeks and then received interactive video game-based exercise in the subsequent 6 weeks. The exercise program consisted of 30-minute sessions 3 times per week for 6 weeks. Outcomes were measured at weeks 0, 6, and 12.
  Interventions: Other: interactive video game-based exercise; Other: no intervention

INTERVENTIONS:
Other: interactive video game-based exercise — Twenty-four patients were randomly allocated to two groups (12 participants per group). Group A received interactive video game-based exercise training for the first 6 weeks, with no intervention in the subsequent 6 weeks. Group B had no intervention for the first 6 weeks and then underwent interactive video game-based exercise training in the subsequent 6 weeks.
Other: no intervention — Twenty-four patients were randomly assigned to two groups (12 participants per group). Group A received interactive video game-based exercise training for the first 6 weeks, with no intervention in the subsequent 6 weeks. Group B had no intervention for the first 6 weeks and then underwent interactive video game-based exercise training in the subsequent 6 weeks.

SUMMARY:
This study assessed the effects of interactive video game-based exercise (IVGB) on balance in persons with Parkinson's disease . Twenty-four patients were randomly allocated to two groups (12 participants per group). Group A underwent IVGB training for the first 6 weeks, with no exercise in the subsequent 6 weeks. Group B had no exercise for the first 6 weeks and then received IVGB training in the subsequent 6 weeks. Both subjective and objective measures were used to determine whether IVGB exercise improves balance function.

DETAILED DESCRIPTION:
The experiments were conducted as a prospective, randomized, single blinded, crossover, 12-week trial. The group A undergoes the IVGB training in the initial 6 weeks (intervention phase), follows by suspended from exercise in the subsequent 6 weeks (control phase). The group B does not received treatment in the first 6 weeks (control phase), and then performs IVGB training in the following 6 weeks (intervention phase). For all participants, The 36-Item Short-Form Health Survey (SF-36), Modified Falls Efficacy Scale (MFES), Berg Balance Scale (BBS), Multidirectional reach test (MDRT) and Maximum step length (MSL) test were assessed at weeks 0, 6, and 12 of the experiment.

ELIGIBILITY:
Inclusion Criteria:

* medical diagnosis of idiopathic Parkinson's Disease
* independent community ambulatory individuals
* capable of giving informed and written consent (Mini-Mental Status Examination (MMSE)>23)

Exclusion Criteria:

* the other neurological conditions such as dementia, and stroke, or if they have arthritis, vision impairment,
* cardiovascular disease that impair walking, or diabetic and uremic individuals, or if they were unable to walk without assistance.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Change of Berg Balance Scale (BBS) | 15 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  Participants perform a series of 14 functional balance tasks, such as maintaining a quiet stance, sitting-to-stand, shifting weight and reaching, turning in place, standing on one leg, and maintaining a tandem stance. The performance of each task is scored on a 5-point ordinal scale (from 0 to 4). A score of 0 denotes the inability of the participant to perform the task, and a score of 4 denotes that the participant can complete the task based on a preset criterion. The highest possible score is 56 . Previous studies have shown that inter-rater and intra-rater reliability of BBS is high in elderly people and stroke patients.

SECONDARY OUTCOMES:
Change of 36-Item Short-Form Health Survey (SF-36) | 15 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  The 8 scales in SF 36 including Physical function (PF), Role-physical (RP), Bodily pain (BP), General health (GH), Vitality (VT), Social Function (SF), Role-Emotional (RE), Mental Health (MH) . Neuromuscular condition is one of the most frequently studied disease with use of SF-36 .
Change of Modified Falls Efficacy Scale (MFES) | 10 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  The MFES is a 14-item rating scale questionnaire that contains the original 10-activity Falls Efficacy Scale and 4 additional activities. Items are rated from 0 (not confident at all) to 10 (completely confident), and the highest possible score is 140.
Change of Multidirectional Reach Test (MDRT) | 10 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  The participants were required to reach in the forward, left and right directions. For the forward-reaching direction, the participants began by raising both arms to the shoulder level. They were then instructed to reach forward as far as they could without moving their feet, while maintaining the end-range position for 3 seconds. A soft measuring tape fixed to the wall was used to measure the start and end positions of the middle finger to measure the reaching distance. The same instructions were provided for the lateral reaching tests, except that the participants lifted only their right or left arm when reaching in the right or left directions, respectively. Three trials were performed in each direction, and the reaching distance was normalized according to the measured foot length.
Change of Maximum Step Length (MSL) test | 10 minutes/session; measured at weeks 0, 6, and 12 of the experiment
  The participants performed the MSL test in the forward, lateral and backward directions. For the forward direction test, the participants assumed the starting position by crossing their arms over their chest. They were then instructed to take a maximum step forward with one leg without moving the other, and then to return to the starting position with a single step.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Lai, MD PhD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical university Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Derived] Yuan RY, Chen SC, Peng CW, Lin YN, Chang YT, Lai CH. Effects of interactive video-game-based exercise on balance in older adults with mild-to-moderate Parkinson's disease. J Neuroeng Rehabil. 2020 Jul 13;17(1):91. doi: 10.1186/s12984-020-00725-y. PMID 32660512